CLINICAL TRIAL: NCT06820281
Title: Acute Metabolic Effects of Tirzepatide in Type 1 Diabetes: a Phase 2 Double Blinded Placebo Controlled Clinical Trial (TIRTLE2)
Brief Title: Acute Metabolic Effects of Tirzepatide in Type 1 Diabetes
Acronym: TIRTLE2
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Garvan Institute of Medical Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: U1111-1316-2752
Record Dates: First submitted 2025-02-06; First posted 2025-02-11 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-01

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Diabetes Mellitus, Type 1; Diabetes Mellitus; Autoimmune Diseases; Incretins; Physiological Effects of Drugs; Tirzepatide; Glucose Metabolism Disorders; Metabolic Diseases; Endocrine System Diseases; Overnutrition; Insulin Resistance
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus; Autoimmune Diseases; Glucose Metabolism Disorders; Metabolic Diseases; Endocrine System Diseases; Overnutrition; Insulin Resistance | interventions — Tirzepatide; Saline Solution

STUDY DESIGN:
Intervention Model Description: Parallel assignment, 1:1 randomization
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Tirzepatide 2.5mg weekly (Experimental): Administered subcutaneously.
  Interventions: Drug: Tirzepatide 2.5mg weekly
- Placebo (Placebo Comparator): Administered subcutaneously.
  Interventions: Drug: Placebo injection (normal saline)

INTERVENTIONS:
Drug: Tirzepatide 2.5mg weekly — Tirzepatide 2.5 mg/0.5 mL solution for injection vial or pre-filled pen. Each vial/ pre-filled pen contains tirzepatide 2.5 mg in 0.5 mL solution (2.5mg in 0.6mL if Kwikpen)
  Tirzepatide will be administered by drawing up into a syringe, then administering by subcutaneous injection weekly by study nurses.
  Arms: Tirzepatide 2.5mg weekly
Drug: Placebo injection (normal saline) — Placebo will be given as 0.5mL normal saline (if comparator against vial or pre-filled pen), or 0.6mL (if comparator against Mounjaro Kwikpen), drawn up into a syringe and administered by subcutaneous injection weekly by study nurses.
  Arms: Placebo

SUMMARY:
This study will examine the effects of Tirzepatide (TZP), a glucagon-like peptide 1 (GLP1) - gastric inhibitory peptide (GIP) co-agonist, on metabolism in type 1 diabetes (T1D). Research participants with T1D will undergo measures of insulin sensitivity, and hormone levels post-meal, post-hypoglycemia and during the overnight period. These measures will be performed prior to, and after 6 weeks of treatment with TZP or placebo.

DETAILED DESCRIPTION:
TIRTLE2 is a phase 2 double-blinded placebo-controlled mechanistic clinical trial that extends upon the findings of TIRTLE1, a phase 2 double-blinded placebo-controlled trial (TZP 5.0mg vs placebo over 12 weeks) in T1D (trial registration: ACTRN12624000111572).

TIRTLE2 is a designed to determine whether TZP can 1) improve whole body insulin sensitivity, 2) reduce prandial glucagon secretion, 3) impacts lipolysis and growth hormone secretion overnight, and 4) determine if TZP can maintain the glucagon response to hypoglycemia. The acute effects of TZP on metabolism will be assessed after 6 weeks, to limit the degree of weight loss (indicating a role for TZP on improving metabolic physiology in T1D, beyond weight management in T1D).

To address these research aims, a single comprehensive clinical trial will be performed in 44 participants with T1D, who will receive a weekly injection of TZP 2.5mg or placebo for 6 weeks. A short treatment duration was chosen to assess if TZP offers T1D-specific benefits prior to significant weight loss.

TIRTLE2 will employ the 'gold standard' hyperinsulinemic-euglycemic and hypoglycemic clamps, in conjunction with complementary analyses of the effects of TZP on metabolism across multiple physiological states. This mechanistic study will define mechanisms by which GLP1-GIP co-agonism may uniquely provide clinical benefits in T1D during the fasting and fed states, and during hypoglycemia.

ELIGIBILITY:
Inclusion Criteria:

* age 18-65 years
* BMI ≥ 27 kg/m2
* HbA1c ≤ 9.0%
* insulin delivery using an automated insulin delivery system
* at least 2 years since diagnosis of type 1 diabetes

Exclusion Criteria:

* TZP or GLP-1 receptor agonist in last 3 months; metformin or sodium glucose co-transporter 2 (SGLT2) inhibitor in the last 6 weeks; steroids, antipsychotics, immunosuppressants in the last 6 weeks.
* Hypoglycemic unawareness or severe hypoglycemia last 6 months.
* History of seizure disorder.
* History of weight loss surgery.
* eGFR <60 mL/min/1.73 m2.
* Liver disease (known cirrhosis, LFTs > 3x upper limit of normal).
* Active malignancy.
* Pregnant, breastfeeding, planning pregnancy within 6 months, or not using adequate contraception.
* History of cardiovascular disease, or coronary event or stroke in last 3 months
* Hemoglobin level < 13.5 g/dL in men, < 12.0 g/dL in women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Whole-body insulin sensitivity | 6 weeks
  Change in insulin sensitivity from baseline, assessed using the hyperinsulinemic-euglycemic clamp (60 mU/m2/min)

SECONDARY OUTCOMES:
Prandial glucagon secretion | 6 weeks
  Change from baseline glucagon area under the curve (AUC) during mixed meal tolerance test (MMTT)
Glucagon response to hypoglycemia | 6 weeks
  Change from baseline glucagon AUC after glucose nadir as measured during the hyperinsulinemic hypoglycemic clamp
% Time level 2 hypoglycemia | 6 weeks
  Change from baseline % time level 2 hypoglycemia (defined by glucose < 54 mg/dL [<3.0 mmol/L]) as measured by continuous glucose monitoring
% Time level 1 hypoglycemia | 6 weeks
  Change from baseline % time level 1 hypoglycemia (defined by glucose < 70 mg/dL [3.9 mmol/L] and ≥ 54 mg/dL [3.0 mmol/L]) as measured by continuous glucose monitoring
Resting energy expenditure (REE) | 6 weeks
  Change from baseline REE as measured by indirect calorimetry
Overnight growth hormone curve | 6 weeks
  Change from baseline growth hormone area under the curve (AUC) as measured overnight blood samples
Overnight free-fatty acids (FFA) curve | 6 weeks
  Change from baseline FFA under the curve (AUC) as measured overnight blood samples
Total daily insulin dose | 6 weeks
  Change from baseline total daily insulin dose as measured by pump record
Total daily basal insulin dose | 6 weeks
  Change from baseline total daily basal insulin dose as measured by pump record
Total daily bolus insulin dose | 6 weeks
  Change from baseline total daily bolus insulin dose as measured by pump record
% Time in Range (TIR) | 6 weeks
  Change from baseline %TIR (defined by % readings between 70mg/dL - 180 mg/dL [3.9 - 10.0 mmol/L]) as measured by continuous glucose monitoring
% Time Below Range (TBR) | 6 weeks
  Change from baseline %TBR (defined by % readings below 70mg/dL [3.9mmol/L]) as measured by continuous glucose monitoring
% Time level 1 hyperglycemia | 6 weeks
  Change from baseline % time level 1 hyperglycemia (defined by glucose > 180 mg/dL [10 mmol/L] and glucose ≤ 250 mg/dL [13.9 mmol/L]) as measured by continuous glucose monitoring
% Time level 2 hyperglycemia | 6 weeks
  Change from baseline % time level 1 hyperglycemia (defined by glucose > 250 mg/dL [13.9 mmol/L])) as measured by continuous glucose monitoring
Glycemic variability | 6 weeks
  Change from glycemic variability as measured by continuous glucose monitoring
Gastric emptying | 6 weeks
  Change from baseline gastric emptying during the mixed meal tolerance test (MMTT) assessed using radiolabelled isotope and breath sampling

OTHER OUTCOMES:
Diabetes Treatment Satisfaction | 6 weeks
  Change from baseline diabetes treatment satisfaction, as measured by questionnaire (DTSQ)
Metanephrine response to hypoglycemia | 6 weeks
  Change from baseline peak metanephrine after glucose nadir as measured during the hyperinsulinemic hypoglycemic clamp
Normetanephrine response to hypoglycemia | 6 weeks
  Change from baseline peak normetanephrine after glucose nadir as measured during the hyperinsulinemic hypoglycemic clamp
Growth hormone response to hypoglycemia | 6 weeks
  Change from baseline peak growth hormone after glucose nadir as measured during the hyperinsulinemic hypoglycemic clamp
Cortisol response to hypoglycemia | 6 weeks
  Change from baseline peak cortisol after glucose nadir as measured during the hyperinsulinemic hypoglycemic clamp
Glucose requirement to correct hypoglycemia | 6 weeks
  Change from baseline glucose infusion requirement after glucose nadir to correct hypoglycemia during the hyperinsulinemic hypoglycemic clamp
Body weight | 6 weeks
  Change from baseline body weight as measured by scale
% fat free mass | 6 weeks
  Change from baseline % fat free mass as measured by air displacement plethysmography
% fat mass | 6 weeks
  Change from baseline % fat mass as measured by air displacement plethysmography
Lipid profile | 6 weeks
  Change from baseline lipid profile as measured by blood assay
Systolic blood pressure | 6 weeks
  Change from baseline systolic blood pressure as measured by digital sphygmomanometer
Diastolic blood pressure | 6 weeks
  Change from baseline diastolic blood pressure as measured by digital sphygmomanometer
Arterial stiffness | 6 weeks
  Change from baseline arterial stiffness as measured by Augmentation index (AIx) by radial artery tonometry
Arterial stiffness | 6 weeks
  Change from baseline arterial stiffness as measured by carotid femoral pulse-wave velocity (cfPWV)
Prandial GLP1 secretion | 6 weeks
  Change from baseline GLP1 area under the curve (AUC) during mixed meal tolerance test (MMTT)
Prandial GIP secretion | 6 weeks
  Change from baseline GIP area under the curve (AUC) during mixed meal tolerance test (MMTT)
Fasting glucagon | 6 weeks
  Change from baseline fasting glucagon level as measured by blood assay.
Fasting GLP1 | 6 weeks
  Change from baseline fasting GLP1 as measured by blood assay
Fasting GIP | 6 weeks
  Change from baseline fasting GIP as measured by blood assay
Supraclavicular temperature profile | 6 weeks
  Change from baseline supraclavicular temperature profile as measured by temperature sensor
Diet composition | 6 weeks
  Change from baseline diet composition as measured by self-reported diet diary entries
Growth differentiation factor 15 (GDF15) | 6 weeks
  Change from baseline fasting GDF15 as measured by blood assay
Fasting liver function tests | 6 weeks
  Change from baseline fasting liver function tests as measured by blood assay
Pulse rate | 6 weeks
  Change from baseline pulse rate as measured by digital sphygmomanometer
C-terminal telopeptide of type 1 collagen | 6 weeks
  Change from baseline C-terminal telopeptide of type 1 collagen (CTX) as measured by blood assay
Procollagen type 1 N-terminal propeptide | 6 weeks
  Change from baseline procollagen type 1 N-terminal propeptide (P1NP) as measured by by blood assay
HbA1c | 6 weeks
  Change from baseline HbA1c as measured by blood assay.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer R Snaith, MD PHD, Principal Investigator — Victor Chang Cardiac Research Institute; Jerry R Greenfield, MD PHD, Study Director — Victor Chang Cardiac Research Institute
Locations (1):
- Garvan Institute of Medical Research, Sydney, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: Yes
Data from these analyses can be made available upon the condition of compliance with institutional review board restrictions and a data sharing agreement with the project sponsor. We encourage researchers who propose use of study data to contact the study PI.